CLINICAL TRIAL: NCT01364012
Title: A Randomized, Double-blinded, Placebo-controlled, Multicenter Phase III Study Comparing Bevacizumab Plus Carboplatin/Paclitaxel Versus Placebo Plus Carboplatin/Paclitaxel in Patients With Advanced or Recurrent Non-Squamous Non-Small Cell Lung Cancer Who Have Not Received Prior Chemotherapy For Advanced Disease
Brief Title: A Study of Bevacizumab Versus Placebo in Combination With Carboplatin/Paclitaxel in Participants With Advanced or Recurrent Non-Squamous Non-Small Cell Lung Cancer Who Have Not Received Previous Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YO25404
Record Dates: First submitted 2011-05-27; First posted 2011-06-02 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Bevacizumab + Paclitaxel/Carboplatin (Experimental): Participants will receive bevacizumab on Day 1 of each 3-week cycle in combination with paclitaxel and carboplatin for the first 6 treatment cycles (cycle length = 21 days). Participants will continue to receive bevacizumab on Day 1 of each 3-week cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Bevacizumab; Drug: Carboplatin; Drug: Paclitaxel
- Placebo + Paclitaxel/Carboplatin (Active Comparator): Participants will receive bevacizumab matching placebo on Day 1 of each 3-week cycle in combination with paclitaxel and carboplatin for the first 6 treatment cycles (cycle length = 21 days). Participants will continue to receive bevacizumab matching placebo on Day 1 of each 3-week cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab will be administered at 15 mg/kg IV on Day 1 of each 3-week cycle until disease progression or unacceptable toxicity.
  Other Names: Avastin
  Arms: Bevacizumab + Paclitaxel/Carboplatin
Drug: Carboplatin — Carboplatin will be administered at area under the plasma concentration-time curve (AUC) 6.0 IV on Day 1 of each 3-week cycle, up to 6 cycles.
Drug: Paclitaxel — Paclitaxel will be administered at 175 milligrams per square meter (mg/m^2) IV on Day 1 of each 3-week cycle, up to 6 cycles.
Drug: Placebo — Bevacizumab matching placebo will be administered IV on Day 1 of each 3-week cycle until disease progression or unacceptable toxicity.
  Arms: Placebo + Paclitaxel/Carboplatin

SUMMARY:
This randomized, double-blind, placebo-controlled study will evaluate the efficacy and safety of bevacizumab (Avastin) versus placebo in combination with carboplatin/paclitaxel in participants with advanced or recurrent non-squamous non-small cell lung cancer who have not received prior chemotherapy for advanced disease. Participants will be randomized to receive either bevacizumab 15 milligrams per kilogram (mg/kg) intravenously (IV) or placebo on Day 1 of each 3 week cycle, plus up to 6 cycles of carboplatin/paclitaxel. Anticipated time on study treatment is until disease progression or unacceptable toxicity occurs. After progression, participants in the bevacizumab arm may continue to receive bevacizumab in combination with approved second- and third-line treatment at the discretion of the investigator, up to the third progression.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced (Stage IIIb not amenable for combined modality treatment), metastatic (Stage IV) or recurrent non-squamous non-small cell lung cancer
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Adequate hematological, renal and liver function

Exclusion Criteria:

* Prior chemotherapy or treatment with another systemic anti-cancer agent for the treatment of the participant's current stage of the disease (Stage IIIb, IV or recurrent disease)
* Mixed non-small cell and small cell tumors or mixed adenosquamous carcinomas with a predominant squamous component
* Evidence of tumor invading major blood vessels on imaging
* Central nervous system (CNS) metastases, even if previously treated
* History of hemoptysis in the 3 months prior to enrollment
* History or evidence of inherited bleeding diathesis or coagulopathy
* Uncontrolled hypertension and/or history of hypertensive crisis or hypertensive encephalopathy
* Clinically significant cardiovascular or vascular disease
* Malignancies other than non-small cell lung cancer within 5 years prior to randomization, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, or localized prostate cancer or ductal carcinoma in situ treated surgically with curative intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2011-05-23 (Actual); Primary Completion 2013-01-27 (Actual); Study Completion 2017-08-17 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) as Assessed Using Response Evaluation Criteria in Solid Tumors Version 1.0 (RECIST v1.0) Criteria | Baseline up to death or disease progression, whichever occurs first (up to approximately 20 months)

SECONDARY OUTCOMES:
Overall Survival (OS) | Baseline up to death (up to approximately 35 months)
Percentage of Participants Who are Alive at Year 1 | Year 1
Percentage of Participants With Objective Response of Complete Response (CR) or Partial Response (PR) as Assessed Using RECIST v1.0 Criteria | Baseline up to death or disease progression, whichever occurs first (up to approximately 35 months)
Duration of Response as Assessed Using RECIST v1.0 Criteria | Baseline up to death or disease progression, whichever occurs first (up to approximately 35 months)
Percentage of Participants With Adverse Events | From baseline up to approximately 35 months
PFS as Assessed Using RECIST v1.0 Criteria in Subgroups Defined by Vascular Endothelial Growth Factor-A (VEGF-A) High/Low Level Expression at Baseline | Baseline up to death or disease progression, whichever occurs first (up to approximately 35 months)
PFS as Assessed Using RECIST v1.0 Criteria in Subgroups Defined by Vascular Endothelial Growth Factor Receptor 2 (VEGFR-2) High/Low Level Expression at Baseline | Baseline up to death or disease progression, whichever occurs first (up to approximately 35 months)
OS in Subgroups Defined by VEGF-A High/Low Level Expression at Baseline | Baseline up to death (up to approximately 35 months)
OS in Subgroups Defined by VEGFR-2 High/Low Level Expression at Baseline | Baseline up to death (up to approximately 35 months)
Percentage of Participants With Objective Response of CR or PR as Assessed Using RECIST v1.0 Criteria in Subgroups Defined by VEGF-A High/Low Level Expression at Baseline | Baseline up to death or disease progression, whichever occurs first (up to approximately 35 months)
Percentage of Participants With Objective Response of CR or PR as Assessed Using RECIST v1.0 Criteria in Subgroups Defined by VEGFR-2 High/Low Level Expression at Baseline | Baseline up to death or disease progression, whichever occurs first (up to approximately 35 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- China (17):
  - The Affiliated Hospital of Military Medical Sciences(The 307th Hospital of Chinese PLA), Beijing
  - Beijing Cancer Hospital, Beijing
  - Beijing Hospital of Ministry of Health; Hematology, Beijing
  - General Hospital of Chinese PLA; Department of Hematology, Beijing
  - Beijing Chest Hospital; Oncology Department, Beijing
  - The Second Xiangya Hospital of Central South University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - Guangdong General Hospital, Guangzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jiangsu Cancer Hospital, Nanjing
  - Guangxi Cancer Hospital of Guangxi Medical University, Nanning
  - Shanghai chest hospital, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Cancer Hospital of Shantou University Medical College, Shantou

REFERENCES:
- [Derived] Zhou C, Wu YL, Chen G, Liu X, Zhu Y, Lu S, Feng J, He J, Han B, Wang J, Jiang G, Hu C, Zhang H, Cheng G, Song X, Lu Y, Pan H, Zheng W, Yin AY. BEYOND: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase III Study of First-Line Carboplatin/Paclitaxel Plus Bevacizumab or Placebo in Chinese Patients With Advanced or Recurrent Nonsquamous Non-Small-Cell Lung Cancer. J Clin Oncol. 2015 Jul 1;33(19):2197-204. doi: 10.1200/JCO.2014.59.4424. Epub 2015 May 26. PMID 26014294